CLINICAL TRIAL: NCT02660710
Title: LCCC 1335: A Single-Arm Phase I/II Clinical Trial of Rituximab Plus CHOP Chemotherapy for Diffuse Large B-cell Lymphoma in Malawi
Brief Title: Rituximab Plus CHOP Chemotherapy for Diffuse Large B-cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH); National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 1335; K01TW009488 (NIH); R21CA180815 (NIH)
Record Dates: First submitted 2016-01-17; First posted 2016-01-21 (Estimated); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Diffuse Large B-cell Lymphoma; HIV
Keywords: single arm phase 2; safety and efficacy; R-CHOP
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — R-CHOP protocol; Rituximab; Reditux

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- R-CHOP (Experimental): We will enroll 40 adult patients age 18-60 years (20 HIV-infected with CD4 count ≥ 100 cells/µL, 20 HIV-uninfected) who will receive a maximum of 6-8 cycles of rituximab plus cyclophosphamide, doxorubicin, vincristine, prednisone (R-CHOP) over 18-24 weeks
  Interventions: Drug: R-CHOP

INTERVENTIONS:
Drug: R-CHOP — maximum of 6-8 cycles of R-CHOP over 18-24 weeks
  Other Names: Indian generic biosimilar for rituximab, Reditux™

SUMMARY:
The purpose of this study is to establish the safety of rituximab plus cyclophosphamide, doxorubicin, vincristine,prednisone (R-CHOP) in HIV-infected and HIV-uninfected diffuse large B-cell lymphoma (DLBCL) patients in Malawi.

DETAILED DESCRIPTION:
The study is a single-center, non-randomized phase II clinical trial of R-CHOP for CD20-positive DLBCL, using the Indian generic biosimilar for rituximab, Reditux™. The investigators will enroll 40 adult patients age 18-60 years (20 HIV-infected with CD4 count ≥ 100 cells/µL, 20 HIV-uninfected) who will receive a maximum of 6-8 cycles of R-CHOP over 18-24 weeks. The primary goal of this study is to establish the safety of R-CHOP in the Malawi population.

Secondary objectives of the study include estimates of complete response (CR) rates, progression-free survival (PFS), and overall survival (OS). In addition, quality of life, costs of care, study patient characteristics, clinical outcomes and other published data from the region will be collected and used to evaluate the cost-effectiveness of R-CHOP. If the investigators' study supports incorporating rituximab into treatment regimens in sub-Saharan Africa, this strategy can be examined in larger trials, and provide momentum to increase access to modern cancer medicines globally.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained and signed. Age 18-60 years. ECOG performance status (PS) 0-2. Histologically confirmed CD20-positive DLBCL, any stage, bulky or nonbulky disease.
* No prior treatment for lymphoma. Willing to have documentation of HIV status. CD4 count ≥ 100 cells/µL if HIV-infected. Measurable disease by physical exam.
* Adequate bone marrow renal and hepatic function as evidenced by the following:

  * Absolute neutrophil count (ANC) ≥ 1,000/µL
  * Platelet count ≥ 100,000/µL
  * Creatinine ≤ 1.5 mg/dL
  * Total bilirubin ≤ 2 mg/dL (unless directly attributable to lymphoma)
* Able to understand and comply with protocol requirements for the entire length of the study.
* Willing to reside <50 kilometers from Kamuzu Central Hospital (KCH) until chemotherapy completion.
* Negative urine B-HCG in women of child-bearing potential within 7 days prior to start of treatment.
* Fertile patients must use effective contraception (condom or other barrier methods, oral contraceptives, implantable contraceptives, intrauterine devices) during and for six months after completion of treatment.

Exclusion Criteria

* Pregnant or nursing. Central nervous system (CNS) involvement by lymphoma (clinically or cytologically confirmed).
* Receiving other anti-cancer or investigational therapy during study treatment, apart from those agents specified in the study protocol.
* Known cardiac disease including any of the following:

  * New York Heart Association (NYHA) Grade II or greater congestive heart failure
  * History of myocardial infarction or unstable angina within 6 months prior to Day 1
  * History of stroke or transient ischemic attack within 6 months prior to Day 1
* Second active malignancy requiring systemic therapy.
* Hepatitis B virus (HBV) surface-antigen positive unless receiving both tenofovir and lamivudine as part of antiretroviral therapy if HIV-infected.
* Other serious, ongoing, non-malignant disease or infection that would in the opinion of the site investigator compromise other protocol objectives.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2016-03; Primary Completion 2021-07-22 (Actual); Study Completion 2022-07-22 (Actual)

PRIMARY OUTCOMES:
Number of DLBCL patients receiving R-CHOP who experience NCI grade 3 or 4 non-hematologic toxicities | 5 years
  Safety will be assessed by grading toxicity events according to NCI Common Terminology Criteria for Adverse Events version 4.0 (NCI CTCAEv4) other than for hypersensitivity reactions to rituximab. Toxicities will be assessed, graded and documented by investigators at each clinic visit, and then tabulated.
Number of patients who experience treatment-related death over a course of six cycles | 5 years

SECONDARY OUTCOMES:
Number of DLBCL patients by HIV status receiving R-CHOP who experience grade 3 or 4 non-hematologic toxicities over a course of six cycles | 5 years
Number of patients receiving ≥ 90% of the prescribed doses of doxorubicin and cyclophosphamide, respectively among DLBCL patients in Malawi with HIV infection | 24 months
Number of patients receiving ≥ 90% of the prescribed doses of doxorubicin and cyclophosphamide, respectively among DLBCL patients in Malawi without HIV infection | 24 months
Number of patients with progression free survival with R-CHOP administered | 5 years
Number of patients with overall survival with R-CHOP administered | 5 years
Number of patients with complete response rates with R-CHOP administered | 24 months
Number of years from treatment initiation until disease progression or death. | 5 years
  Questionnaire - health-related quality of life (via the EORTC QLQ-C30) among DLBCL patients in Malawi overall and with and without HIV infection receiving R-CHOP
Number of years gained after rituximab plus CHOP chemotherapy administered | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Painschab, MD, Principal Investigator — University of North Carolina
Locations (1):
- UNC Project, Lighthouse Trust, Lilongwe, Malawi

REFERENCES:
- [Derived] Kimani S, Painschab MS, Kaimila B, Kasonkanji E, Zuze T, Tomoka T, Mulenga M, Nyasosela R, Chikasema M, Mtangwanika A, Chawinga M, Mhango W, Nicholas S, Chimzimu F, Kampani C, Krysiak R, Lilly A, Randall C, Seguin R, Westmoreland KD, Montgomery ND, Fedoriw Y, Gopal S. Safety and efficacy of rituximab in patients with diffuse large B-cell lymphoma in Malawi: a prospective, single-arm, non-randomised phase 1/2 clinical trial. Lancet Glob Health. 2021 Jul;9(7):e1008-e1016. doi: 10.1016/S2214-109X(21)00181-9. Epub 2021 May 19. PMID 34022150